CLINICAL TRIAL: NCT05984966
Title: Supported Employment to Create a Community Culture of COVID-19 Rapid Testing Among People Who Inject Drugs: PeerConnect2Test
Brief Title: Supported Employment COVID-19 Rapid Testing for PWID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000657
Record Dates: First submitted 2023-02-28; First posted 2023-08-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Employment, Supported

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supported Employment (Experimental): Supported employment program (Peer Connect2Test) for people who inject drugs to provide SARS-CoV-2 rapid tests to others in their networks
  Interventions: Behavioral: Supported Employment

INTERVENTIONS:
Behavioral: Supported Employment — PeerC2T is part of a supported employment program where PWID are trained and supported to provide PWID with job skills to be able to act as Peer Health Worker to facilitate distribution of rapid SARS-CoV-2 testing to other PWID. The effect of the training on the Peer Health Worker themself will be evaluated (Aim 1). In addition, in Aim 2 they will distribute the rapid test kits in places of residence such as tents, shelters, apartments, trailers, or houses or locations where other PWID frequently engage with services such as syringe exchange. The kit is the BinaxNOW COVID-19 Antigen Self Test, which is approved to be used as a lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2. PWID community members will be offered a free test kit, and the Peer Health Worker will record whether the community member elected to take the test (yes/no), and they will also collect administrative demographic data on the PWID.
  Other Names: Peer Connect2Test

SUMMARY:
This community-engaged project aims to improve the accessibility of rapid tests through a supported employment program for people who inject drugs (PWID). The program is called Peer Connect2Test (PeerC2T). PWID will be recruited by a community partner who provides syringe exchange services. PWID will the trained by the community partner to become peer health workers (PHW) to distribute SARS-CoV-2 rapid tests to other PWID. Investigators expect that PeerC2T will improve knowledge, self-efficacy, and health behaviors among PHW (Aim 1). The study will use the RE-AIM framework in Aims 2 and 3 to evaluate whether PeerC2T improves SARS-CoV-2 testing uptake among other PWID (RE; Aim 2), and identify intervention considerations (AIM; Aim 3). The overall goal of this project is develop a transformative community-driven intervention in partnership with a community partner to promote widespread access to rapid testing among PWID.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older, understand English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative semi-structured interview with PWID Peer Health Worker | 3 months post intervention involvement
  Includes:(a) provided participant with purpose and meaning; (b) helped them create more meaningful social relationships; (c) provided opportunities for engaging with society in a positive way; (d) helped them feel competent and capable; and (e) facilitated optimism about the future. Coded using NVivo text-analysis software.
Change in Self-efficacy of PWID Peer Health Worker | Change from Baseline Self-efficacy at 3 months
  To test Aim 1 using qualitative data, we will develop self-efficacy items based on skills taught in the supported employment training 5-point response option (1 = Strongly disagree, 5 = strongly agree).
Change in Behavioral Intentions of Peer Health Worker | Change from Baseline Behavior at 3 months
  To test Aim 1, we will adapt questions from the Preventative Medicine Attitudes and Activities Questionnaire, and using the same response option, reframe the items based on how often they intend to engage in the behavior. We will develop the knowledge items based on skills taught in the training. Higher scores indicate greater behavioral intentions.
Change in Flourishing Scale (Well-Being) | Change from Baseline Flourishing (well-being) at 3 months
  To test Aim 1, we will use an 8-item summary measure of self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism. Questions pertain to experiences over the past 4-weeks (e.g., My social relationships are supportive and rewarding, I am engaged and interested in my daily activities) and responses are indicated on a 7-point scale (1 = Strongly disagree, 7 = Strongly agree). The possible range of scores is from 8 (lowest possible) to 56 (highest PWB possible). A high score represents a person with many psychological resources and strengths
Percent of people who inject drugs who agree to testing for COVID-19 | through study completion, an average of 1 year
  Peer Health Workers will offer a rapid test to 1000 PWID. The percent of PWID who agree to take the test serves as this measure for Aim 2a.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data with the RADx-UP Data Coordination Center at Duke University. Data will be de-identified and available to other researchers for further use.
Supporting Information: Study Protocol, ICF
Time Frame: Upon study completion. Timeframe available determined by the National Institutes of Health.
URL: https://radx-up.org/research/cdes/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT05984966/Prot_ICF_000.pdf